CLINICAL TRIAL: NCT06779071
Title: A Multicenter, Randomized, Double-blinded, Active-controlled, Non-inferiority, Pivotal Clinical Trial to Evaluate the Efficacy and Safety in Pain Reduction After NPNP-001 Application in the Knee Joint of Patients with Knee Osteoarthritis
Brief Title: Pivotal Clinical Trial to Evaluate the Efficacy and Safety After NPNP-001 Application in Patients with Knee Osteoarthritis.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaResearch Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-NPNP001-P3-02
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: Polynucleotide sodium; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPNP-001 (Experimental)
  Interventions: Device: NPNP-001
- Conjuran (Active Comparator)
  Interventions: Device: Conjuran

INTERVENTIONS:
Device: NPNP-001 — Description: NPNP-001 2ml per injection, once a week for 3 injections. Placebo(saline) 2ml per injection, once a week for 2 injections.
  Other Names: Polynucleotide sodium (PN)
  Arms: NPNP-001
Device: Conjuran — Description: Conjuran 2ml per injection, once a week for 5 injections.
  Other Names: Polynucleotide sodium (PN)
  Arms: Conjuran

SUMMARY:
This study was designed to demonstrate non-inferiority and safety in pain reduction after NPNP-001 application in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 40 years or older as of the date of written consent
2. Patients diagnosed with unilateral or bilateral knee osteoarthritis according to the American College of Rheumatology (ACR) clinical diagnostic criteria, experiencing knee joint pain, and meeting at least three of the following conditions:

   * Age > 50 years
   * Morning stiffness < 30 minutes
   * Crepitus
   * Bony tenderness
   * Bony enlargement
   * No palpable warmth of the synovium
3. At least one knee joint with a Weight-Bearing Pain (100 mm-VAS) score ≥ 40 mm, measured at the screening visit
4. X-ray results from within 6 months prior to screening or at the screening visit indicating that the target lesion of knee osteoarthritis corresponds to Kellgren Lawrence Grade 1 to 3.
5. Patients with knee osteoarthritis who have not responded to conservative treatments such as pharmacotherapy or physical therapy for at least 3 months prior to screening.
6. Patients who can adequately understand and complete the efficacy assessment questionnaires.
7. Patients who voluntarily agree to the informed consent form after receiving an explanation of the purpose, methods, and effects of the clinical trial.
8. Patients who agree to refrain from using any pharmacotherapy for knee osteoarthritis other than the rescue medication during the clinical trial period.
9. Patients who are able to undergo allergy testing (skin prick test).

Exclusion Criteria:

1. Patients with a Body Mass Index (BMI) ≥ 35 kg/m² at screening.
2. Patients with rheumatoid arthritis or other types of arthritis such as traumatic, metabolic, etc.
3. Patients with conditions that are deemed likely to affect the efficacy and safety assessment of this clinical trial (however, those who are considered eligible by the investigator may be enrolled):

   * Patients with severe painful conditions such as septic arthritis, autoimmune diseases, gout, recurrent pseudogout, Paget's disease, etc.(e.g. Sudeck's atrophy, herniated discs, etc.), as well as those with joint fractures, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondrosis, genetic diseases (hyperkinesis, etc.), collagen gene abnormalities
   * Patients with hemorrhagic disorders, hemostatic disorders, CNS diseases, cancer, AIDS, heart disease, kidney disease, uncontrolled diabetes and hypertension, severe medical or psychiatric conditions, and patients with hypersensitivity to local anesthetics.
4. Patients with severe osteoarthritis symptoms in other joints (e.g., hip joint) that may affect pain assessment in the knee joint (polyarticular joint pain).
5. Patients with skin abnormalities at the injection site that may affect invasive procedures, such as infections or skin diseases.
6. Patients who have received the following medications prior to screening:

   A. Patients who have received sodium polynucleotide and/or hyaluronic acid(HA) injections into the target knee joint within 6 months prior to screening.

   B. Patients who have received steroid injections into the target knee joint within 3 months prior to screening.

   C. Patients who have used systemic steroids within 1 month prior to screening (topical and inhaled steroids are excluded).

   D. Patients who have received cell therapy or gene therapy into the target knee joint prior to screening.
7. Patients with severe joint effusion confirmed through tests such as the patellar tap test.
8. Patients who have undergone surgical procedures on the target knee joint or cartilage regeneration surgeries (such as microfracture, autologous chondrocyte implantation, etc.) within 6 months prior to screening (however, patients with surgical history on the opposite knee or hip joints will only be excluded if it is likely to impact the clinical evaluation of the target knee joint).
9. Patients with a history of knee joint replacement surgery in the target joint.
10. Patients who have taken anticoagulants (including warfarin, NOACs [Non-vitamin K Oral Anti-Coagulants], antiplatelet agents [aspirin, clopidogrel; however, low-dose aspirin [100 mg, maximum 300 mg/day] is excluded], thrombolytics [urokinase, alteplase, etc.]) within 2 weeks prior to the application of the investigational device.
11. Patients with a positive allergy test (skin prick test) result for the investigational device conducted at screening or those with hypersensitivity to components of the investigational device used in this clinical trial (including allergies to salmon, shrimp, and crab).
12. Patients who have participated in another clinical trial and received investigational products or medical devices within 6 months prior to screening.
13. Pregnant or breastfeeding women, women of childbearing potential who plan to become pregnant during the clinical trial period and for 3 months after, or men who do not intend to use appropriate contraceptive methods*.

    * Hormonal contraceptives, intrauterine devices (such as Implanon), dual barrier methods (using both male condoms and cervical caps), and sterilization procedures (vasectomy, bilateral tubal ligation, etc.).
14. Patients with knee joint instability.
15. Patients who are expected to start medication for depression or anxiety disorders during the clinical trial period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 260 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Weight-bearing pain (WBP) - 100mm visual analogue scale (VAS) | 20 weeks
  Weight-bearing pain (WBP) - 100mm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Change from baseline of Weight-bearing pain (WBP) - 100mm visual analogue scale (VAS) | 3, 4, 8, 28 weeks
  Weight-bearing pain - 100mm visual analogue scale (VAS)
Change from baseline of Rest pain - 100mm visual analogue scale (VAS) | 3, 4, 8, 20, 28 weeks
  Rest pain - 100mm visual analogue scale (VAS)
Change from baseline of Motion pain - 100mm visual analogue scale (VAS) | 3, 4, 8, 20, 28 weeks
  Motion pain - 100mm visual analogue scale (VAS)
Change from baseline of Patient Global Assessment (PGA) - 100mm visual analogue scale (VAS) | 3, 4, 8, 20, 28 weeks
  Change from baseline of Patient Global Assessment (PGA) - 100mm visual analogue scale (VAS)
Change from baseline of Investigator Global Assessment (IGA) - 100mm visual analogue scale (VAS) | 3, 4, 8, 20, 28 weeks
  Change from baseline of Investigator Global Assessment (IGA) - 100mm visual analogue scale (VAS)
Change from baseline of WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) total score and individual score evaluation (Pain, Function, Stiffness) | 3, 4, 8, 20, 28 weeks
  Change from baseline of WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) total score and individual score evaluation (pain, stiffness, physical function, ) - WOMAC-Likert Assessment (5-point Likert scale: none(0), mild(1), moderate(2), severe(3), and extreme(4)).
  1. The pain subscale consists of 5 questions. The sum of all items of pain subscale ranges from 0 to 20. A higher score indicates worse pain.
  2. The stiffness subscale consists of 2 questions. The sum of all items of the stiffness subscale ranges from 0 to 8. A higher score on the stiffness indicates worse articular function.
  3. The physical function Subscale consists of 17 questions. The sum of all items of the physical function subscale ranges from 0 to 68. A higher score indicates worse functional limitations.
Change from baseline in EQ-5D (EuroQol-5 Dimension Health Questionnaire) Index and EQ VAS(visual analogue scale) assessment to measure quality of life | 3, 4, 8, 20, 28 weeks
  Change from baseline in EQ-5D (EuroQol-5 Dimension Health Questionnaire) Index - 5 Level score and EQ VAS(visual analogue scale) assessment to measure quality of life.
  EQ-5D Index score ranges from 0 to 1, with 0 representing death and 1.0 representing perfect health.
  EQ VAS records participant's self-rated health on a vertical VAS that range from where 0 (worst imaginable) to 100 (best imaginable).
Proportion (%) of participants who took rescue medication at each visit following the application of the investigational device, and consumption | 0, 1, 2, 3, 4, 8, 20, 28 weeks
  Proportion (%) of participants who took rescue medication at each visit following the application of the investigational device, and consumption
Response Rate following the application of the investigational device | 8, 20, 28 weeks
  Response Rate assessment following the application of the investigational device
Physical assessments at each visit following the application of the investigational device: Swelling, Tenderness on pressure, Range of motion(ROM) | From 0 to 28 weeks
  Physical assessments at each visit following the application of the investigational device: Swelling, Tenderness on pressure, Range of motion(ROM)

OTHER OUTCOMES:
The incidence rate of Pre-treatment adverse events (AEs), treatment-emergent adverse events (TEAEs), Solicited Local AEs and the Serious TEAEs | From 0 to 28 weeks
The incidence rate of abnormal CS at Post-Treatment on Laboratory | From 0 to 28 weeks
The incidence rate of abnormal clinical significance (CS) at Post-Treatment on Electrocardiogram | From 0 to 28 weeks
The incidence rate of abnormal on Physical Examination | From 0 to 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided